CLINICAL TRIAL: NCT03995056
Title: A Randomised Controlled Exercise Intervention in Subjects With Non-alcoholic Fatty Liver Disease
Brief Title: Exercise Study in Subjects With NAFLD
Acronym: BestTreat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Eastern Finland (Other)
Collaborators: European Commission (Other); Leibniz Institute for Natural Product Research and Infection Biology Hans Knöll Institute (Other); Afekta (Unknown); Novogene (Unknown); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Clinical Microbiomics (Unknown); Kuopio Research Institute of Exercise Medicine (Other); Kuopio University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BestTreat
Record Dates: First submitted 2019-06-10; First posted 2019-06-21 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Gastrointestinal Microbiome; Exercise
Keywords: NAFLD; Gut microbiota; high-intensity training
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Motor Activity

STUDY DESIGN:
Intervention Model Description: The study contains two arms. One arm is the control group without any changes in their lifestyle (sedentary lifestyle) and the other arm is the intervention group with a high-intensity interval training. Both groups have no changes in their diets.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control-group (No Intervention): Subjects diagnosed with NAFLD and a sedentary lifestyle will have no changes in their habits and diets.
- Exercise-group (Experimental): This group with diagnosed NAFLD patients will perform a high-intensity aerobic interval exercise training without changing their diets.
  Interventions: Behavioral: high-intensity aerobic interval training

INTERVENTIONS:
Behavioral: high-intensity aerobic interval training — The intervention group will follow a high-intensity interval training protocol on a cycle ergometer for 2 times per week and 1 time an individualised home workout program to have a total exercise amount of 3 hours.
  Leisure time physical activity at baseline as well as during the intervention period will be assessed by Polar Active devices.
  Arms: Exercise-group

SUMMARY:
Non-Alcoholic Fatty Liver Disease is the most common cause of chronic liver diseases. The benign non-alcoholic fatty liver, characterized by excessive fat accumulation, can evolve into non-alcoholic steatohepatitis and liver cancer.

The recommendation nowadays is a lifestyle change with physical exercise and diet to reduce liver fat and improve inflammation. Besides this, a leaky gut and dysbiosis have an impact on the liver, and exercise ameliorates the diversity of gut microbiota and permeability of the intestine.

The aim of this study is to find out a link between exercise and the gut-liver axis regarding the stage of liver adiposity and define exercise-responsive gut microbiome in NAFLD patients

DETAILED DESCRIPTION:
For this 12-week randomised controlled intervention 60 subjects between 18 and 70 years old, diagnosed with NAFLD and body mass index under 35 kg/m2 will be recruited. They will be randomly assigned in a high-intensity aerobic interval training (n=30) and a control group with a sedentary lifestyle (n=30). The intervention group follows a supervised high-intensity aerobic interval training two times per week and additionally, an individualised home workout program to have 3 hours of aerobic training per week. Blood samples, adipose tissue biopsy, 24h-urine and faecal samples will be collected at the baseline, midway (only stool) and at the end of the study. Dietary intake will be analysed at weeks 0, 6, 12.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed NAFLD
* BMI:25 - 35 kg/m^2

Exclusion Criteria:

* acute illness or current evidence of acute or chronic inflammatory or infective diseases
* liver disease (e.g. Wilsons disease/alpha-1-antitrypsin deficiency, Hepatitis B and C, hemochromatosis)
* bleeding disorder, anticoagulation medication
* subjects with diagnosed type 1 diabetes or diagnosed type 2 diabetes with insulin or Glucagon-like peptide-1 agonist treatment
* diagnosed depression and mental illness
* any condition preventing physical activity
* smokers
* alcohol abuse (daily consumption ≥ 30 g for men and ≥ 20 g for women)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-04-19 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-06-18 (Actual)

PRIMARY OUTCOMES:
Changes in liver fat content | 12 weeks (baseline and endpoint)
  Changes in liver fat content by means of magnetic resonance imaging (MRI) /magnetic resonance spectroscopy (MRS)
Gut microbiota changes | 12 weeks (baseline and endpoint)
  Changes in the composition and richness of gut microbiota through metagenomic analyses

SECONDARY OUTCOMES:
Changes in glucose profile | 14 weeks (two weeks preceding the intervention and during the last weeks of the intervention)
  Using Freestyle Libre for 2 weeks before the beginning of the intervention and during the last 2 weeks of the intervention to measure tissue glucose concentrations throughout the day
Changes in protein expression in adipose tissue | 12 weeks (baseline and endpoint)
  To define differences in lipid and glucose metabolism related enzymes, transporters
Changes in low-grade inflammation | 12 weeks (baseline and endpoint)
  Cytokine levels (IL1-RA, TNFα, IL-6, MCP-1, IL-1β, TGF-β, IFN-γ, IL-10) in the blood will be measured by ELISA
The effect on body composition | 12 weeks (baseline and endpoint)
  Body composition will be measured by bioimpedance
Changes in metabolomics | 12 weeks (baseline and endpoint)
  Metabolomics (small molecule intermediates and products of metabolism) in stool, blood and urine will be measured by Liquid chromatography-mass spectrometry (LC-MS)

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Schwab, Prof, Study Director — University of Eastern Finland
Locations (1):
- University of Eastern Finland, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Babu AF, Csader S, Mannisto V, Tauriainen MM, Pentikainen H, Savonen K, Klavus A, Koistinen V, Hanhineva K, Schwab U. Effects of exercise on NAFLD using non-targeted metabolomics in adipose tissue, plasma, urine, and stool. Sci Rep. 2022 Apr 20;12(1):6485. doi: 10.1038/s41598-022-10481-9. PMID 35444259
- [Derived] Csader S, Chen X, Leung H, Mannisto V, Pentikainen H, Tauriainen M-M, Savonen K, El-Nezami H, Schwab U, Panagiotou G. Gut ecological networks reveal associations between bacteria, exercise, and clinical profile in non-alcoholic fatty liver disease patients. mSystems. 2023 Oct 26;8(5):e0022423. doi: 10.1128/msystems.00224-23. Epub 2023 Aug 22. PMID 37606372
- See also: European Union Project: "Building a Gut Microbiome Engineering Toolbox for In-Situ Therapeutic Treatments for Non-alcoholic Fatty Liver Disease" — https://www.besttreat.eu/